CLINICAL TRIAL: NCT03855670
Title: The Role of Physical Activity, Malnutrition and Sarcopenia for the Prediction of Acute Exacerbations and the Evolution of COPD Assessment Test (CAT) in Patients With COPD
Brief Title: The Role of Physical Activity for Acute Exacerbations of COPD
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Maximilian Boesch, Principal Investigator, Cantonal Hospital of St. Gallen
Other Study IDs: EKOS 18/055
Record Dates: First submitted 2019-02-21; First posted 2019-02-27 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators plan to study the association between physical activity, malnutrition and sarcopenia and the occurrence of acute exacerbations of COPD / the evolution of the COPD assessment test (CAT) over 1 year in a telehealthcare cohort of patients with COPD. The investigators hypothesize that malnutrition and/or sarcopenia at baseline and a decline in the fat-free mass index over time is associated with an increased rate of acute exacerbations of COPD and an increased CAT score meaning a higher risk for mortality, morbidity and impairment of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* COPD GOLD stage B or higher
* Written informed consent

Exclusion Criteria:

* Inability to provide written informed consent
* Insufficient knowledge of the trial language

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study cohort will be selected by the Cantonal Hospital St. Gallen (primary care clinic)
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Rate of acute exacerbations of COPD | 12 months
  The primary outcome measure is the rate of acute exacerbations of COPD.

SECONDARY OUTCOMES:
Physical activity | 12 months
  The rate of acute exacerbations of COPD will be correlated to the degree of physical activity measured using an activity tracker in everyday life. The following parameters will be recorded:
  * step count
  * distance travelled
  * calories burned
Fat-free mass index | 12 months
  The rate of acute exacerbations of COPD will be correlated to the fat-free mass index (FFMI) measured at baseline and after 6 and 12 months using bioelectrical impedance analysis (BIA).
Hand grip strenght | 12 months
  The rate of acute exacerbations of COPD will be correlated to the hand grip strength (HGS) measured at baseline and after 6 and 12 months using a dynamometer.
C-reactive protein | 12 months
  The rate of acute exacerbations of COPD will be correlated to the level of serum C-reactive protein (CRP) measured at baseline and after 6 and 12 months.
Total protein | 12 months
  The rate of acute exacerbations of COPD will be correlated to the level of total serum protein measured at baseline and after 6 and 12 months.
Albumin | 12 months
  The rate of acute exacerbations of COPD will be correlated to the level of serum albumin measured at baseline and after 6 and 12 months.
25-OH vitamin D3 | 12 months
  The rate of acute exacerbations of COPD will be correlated to the level of serum 25-OH vitamin D3 measured at baseline and after 6 and 12 months.
COPD assessment test | 12 months
  The rate of acute exacerbations of COPD will be correlated to the COPD assessment test (CAT) score which interrogated on a weekly basis.

CONTACTS AND LOCATIONS:
Locations (1):
- Lung Center, Cantonal Hospital St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lung Center, Cantonal Hospital St.Gallen — http://www.kssg.ch/lungenzentrum
- See also: Cantonal Hospital St. Gallen — http://www.kssg.ch/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT03855670/Prot_SAP_000.pdf